CLINICAL TRIAL: NCT01573689
Title: Bereaving, But Not Alone : the Development and Actualization of a Mutual Aid Group for Children Who Have Lost a Parent.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Valerie Pepin LeBlanc, Social Work Master degree canditate, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VLeblanc - bereaved children
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Mourning,; Grief,; Bereavement.
Keywords: bereaved children, mutual aid group, death, group intervention.
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Group intervention based on mutual aid. — Development of a mutual aid group and his actualization on children between nine and twelve years old who had lost one of their parents.

SUMMARY:
The methodology of this clinical trial is based on the realisation of a group intervention with children who lost a parent. Interviews preintervention and postintervention with participants will be done as well. The purpose of this study is to answer the following question: "What are the benefits for children who are in the process of bereaving a parent to participate in a group work intervention based on the mutual aid model ?". The aim of the research is to explore the benefits for grieving children to participate in an group work intervention based on the mutual aid model. To do so, the research has three distinct objectives : 1) to develop and apply a program of group work interventions for grieving children based on the mutual aid model ; 2) to explore the extent to which participation in the group facilitates changes in the children's discourse about death and the loss of their parents, and 3) to examine, from the children's own perceptive, the possible impact that their participation in the group have on their experience of bereavement.

ELIGIBILITY:
Inclusion Criteria:

* Children between 8 and 12 years old.
* Children who had lost a parent within 3 months and two years before the beginning of the group intervention.

Exclusion Criteria:

* Children who experimented death of his parent by suicide.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Mutual aid group intervention | 8 weeks
  A mutual aid group intervention has been develop to help children who had lost a parent. The activities are based on the theoretical knowledge and needs of grieving children.

SECONDARY OUTCOMES:
Interview before the group intervention | one of 60 minutes
  The interview aim is to know and to understand the experience of each participant about the death of their parent.
Interview after the group intervention | One of 60 minutes
  The aim of this interview is to ask questions about the death and the experience of the children after the end of the group intervention. Through the answers, we will find out about to understanding and the perceptions of the children about the group intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Lumi-Vie, Laval, Quebec, Canada